CLINICAL TRIAL: NCT00927784
Title: The Effect of Intramyocardial Injection of Mesenchymal Precursor Cells on Myocardial Function in LVAD Bridge to Transplant Patients
Brief Title: Effect of Intramyocardial Injection of Mesenchymal Precursor Cells on Heart Function in People Receiving an LVAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrollment has been terminated by the NHLBI for administrative reasons.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Angioblast Systems (Industry)
Responsible Party: Principal Investigator, Annetine Gelijns, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 08-1093; P50HL077096 (NIH)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Mesenchymal Precursor Cells; Left Ventricular Assist Device; LVAD; Congestive Heart Failure; Stem Cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoprotective media alone (Sham Comparator): Participants will receive intramyocardial injections of cryoprotective media alone (placebo).
  Interventions: Drug: Cryoprotective media alone
- Mesenchymal Precursor cells (RevascorTM) (Experimental): Participants will receive intramyocardial injections of low dose (25 million) or higher dose (75 million) MPCs in sequential cohorts.
  Interventions: Biological: Mesenchymal Precursor cells (RevascorTM)

INTERVENTIONS:
Biological: Mesenchymal Precursor cells (RevascorTM) — Participants will receive intramyocardial injections of low dose (25 million) or higher dose (75 million) MPCs (in sequential cohorts).
  Other Names: Mesenchymal Precursor cells; RevascorTM
  Arms: Mesenchymal Precursor cells (RevascorTM)
Drug: Cryoprotective media alone — Participants will receive intramyocardial injections of cryoprotective media (placebo).
  Other Names: placebo
  Arms: Cryoprotective media alone

SUMMARY:
Left ventricular assist devices (LVADs) are one treatment option for people with congestive heart failure. This study will evaluate the safety of injecting mesenchymal precursor cells (MPCs) into the heart during LVAD implantation surgery and examine if injecting MPCs into the heart is effective at improving heart function.

DETAILED DESCRIPTION:
Congestive heart failure is a major health problem and recent estimates indicate that end-stage heart failure with a 2-year mortality rate of 70-80% affects over 60,000 people in the United States each year. For these patients, treatment options are extremely limited. Less than 3,000 heart transplants are available each year because of the severely limited supply of donor hearts. Implantable LVADs, routinely used to support heart transplantation patients who decompensate awaiting a donor heart, were approved by the Food and Drug Administration (FDA) in 2002 for long-term support when heart transplantation is not an option. Few patients, however, achieve sufficient recovery to warrant LVAD explantation and those who do must still contend with ventricular dysfunction. MPCs are normally present in human bone marrow and have been shown to increase the development of blood vessels and new heart muscle cells. The purpose of this study is to determine the safety of injecting MPCs into the heart during LVAD implantation surgery. In addition, this study will examine whether injecting MPCs into the heart is effective at improving heart function.

This study will enroll people who are on the waiting list to receive a donor heart and who are undergoing LVAD implantation surgery. Before the surgery, participants will be randomly assigned to one of two groups. One group of participants will have MPCs injected into their heart during LVAD surgery and the other group of participants will have a control solution (placebo) injected into their heart during the surgery. A portion of heart muscle removed during the surgery will be analyzed. Participants will be monitored by study researchers and blood samples will be collected 12 hours after the LVAD surgery and at 1, 7, 21, 60, and 90 days after the surgery. After that, a medical history review, physical examination, and blood collection will occur every 60 days until a heart transplant occurs or until 12 months after the LVAD implantation, whichever comes first. Heart function testing, which will include an echocardiogram, neuronal function testing, and a 6-minute walk test, will occur 60 and 90 days after the LVAD implantation, and every 2 months thereafter until a heart transplant occurs or until 12 months after the LVAD implantation, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documents
* Age 18 years or older
* If the participant or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after LVAD implantation
* Female participants of childbearing potential must have a negative serum pregnancy test at screening
* Admitted to the clinical center at the time of study entry
* Listed with the United Network for Organ Sharing (UNOS) for heart transplantation
* Clinical indication and accepted candidate for implantation of an FDA- approved LVAD as a bridge to transplantation

Exclusion Criteria:

* Cardiothoracic surgery within 30 days of study entry
* Heart attack within 30 days of study entry
* Prior heart transplantation, left ventricular (LV) reduction surgery, or cardiomyoplasty
* Acute reversible cause of heart failure (e.g., myocarditis, profound hypothyroidism)
* Anticipated requirement for biventricular mechanical support
* Stroke within 30 days of study entry
* Received investigational intervention within 30 days of study entry
* Platelet count less than 100,000/uL within 24 hours of study entry
* Active systemic infection within 48 hours of study entry
* Presence of greater than 10% anti-human leukocyte antigen (HLA) antibody titers with known specificity to the MPC donor HLA antigens
* Known hypersensitivity to dimethyl sulfoxide (DMSO), murine, and/or bovine products
* History of cancer prior to screening (excluding basal cell carcinoma)
* Acute or chronic infectious disease, including but not limited to human immunodeficiency virus (HIV)
* Treatment and/or an incompleted follow-up treatment of any investigational therapy within 6 months of study entry
* Active participation in other research therapy for cardiovascular repair/regeneration
* Prior recipient of stem precursor cell therapy for cardiac repair
* Pregnant or breastfeeding at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ascheim, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Yoshifumi Naka, MD, Principal Investigator — Columbia University
Locations (17):
- United States (17):
  - Sharp Memorial Hospital, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Intermountain Medical Center, Salt Lake City, Utah
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 patients with end-stage CHF and clinical indication for implantation with an FDA-approved LVAD as a bridge-to-transplant were to be enrolled. 40 patients in the low dose cohort(25M)/40 patients in the high dose cohort(75M). Trial enrollment was permanently suspended upon 10 patients enrolled in the low dose cohort due to a change in NIH funding.
Groups:
- Low Dose Cohort: Treatment Group: Intramyocardial injection of study drug (25 million MPC) (Revasacor TM)at the time of LVAD implantation
- Low Dose Cohort: Control Group: Intramyocardial injection of vehicle (50% alpha-MEM/42.5% proFreeze NAO Freezing Medium/7.5%DMSO) at the time of LVAD implantation.
Period: Overall Study
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Started | 8 | 2
Completed | 6 | 2
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 51 (5) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infectious Myocarditis
Time Frame: Measured within 90 days of study entry
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

2. Primary Outcome: Incidence of Myocardial Rupture
Time Frame: Measured within 90 days of study entry
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

3. Primary Outcome: Incidence of Neoplasm
Time Frame: Measured within 90 days of study entry
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

4. Primary Outcome: Incidence of Hypersensitivity Reaction
Time Frame: Measured within 90 days of study entry
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

5. Primary Outcome: Incidence of Immune Sensitization
Time Frame: Measured within 90 days of study entry
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

6. Secondary Outcome: Assessment of LVAD Wean
Description: The secondary endpoints assessed during the LVAD wean include echocardiographic assessments, 6 minute walk, ability to tolerate wean from LVAD support, duration of ability to tolerate wean from LVAD support, and neuronal function.
  Measured at 60 days, 90 days, and every 60 days thereafter following LVAD implantation until heart transplantation or 12 months, whichever comes first
Time Frame: up to 12 months
Population: data not collected
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Study Intervention-related Adverse Events
Description: This includes Device Malfunction-Pump Thrombus-Suspected and Internal Pump Component, Inflow, or Outflow Tract Infection
Time Frame: up to 12 months
Measure: Number; unit: participants
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
participants | 2 | 0

8. Secondary Outcome: Incidence of All Serious Adverse Events
Time Frame: up to 12 months
Measure: Number; unit: events
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 8 | 2
events | 27 | 1

9. Secondary Outcome: Number of Patients Who Experienced Donor-specific HLA Sensitization
Description: Number of patients who experienced donor-specific HLA sensitization post-randomization in each treatment arm.
Time Frame: up to 12 months
Population: Study terminated early. Data not collected or analyzed for this Outcome Measure.
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Myocardial Neovascularization at Time of Explant
Time Frame: up to 12 months
Population: Study terminated early. Data not collected or analyzed for this Outcome Measure
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence of Cardiomyocyte Regeneration at Explant
Time Frame: up to 12 months
Population: Study terminated early. Data not collected or analyzed for this Outcome Measure.
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Incidence of Cell Engraftment and Fate at Explant
Time Frame: up to 12 months
Population: Study terminated early. Data not collected or analyzed for this Outcome Measure.
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Incidence of Survival to Cardiac Transplantation
Time Frame: up to 12 months
Population: Study terminated early. Data not collected or analyzed for this Outcome Measure.
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Continuous from randomization until induction of anesthesia for cardiac transplant or 12 months, whichever comes first.
Description: Adverse events were documented and reported by staff at the study sites as they occurred per the protocol definitions. All adverse events were adjudicated by an Independent Clinical Events Committee (CEC).
Arm/Group | Low Dose Cohort: Treatment Group | Low Dose Cohort: Control Group
Serious Adverse Events (participants affected / at risk) | 8/8 | 1/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Cohort: Treatment Group (N=8) | Low Dose Cohort: Control Group (N=2)
Intra-operative Bleeding (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Major Bleeding (Non-Intra-Operative) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Venous Thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Other Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — elevated INR, epistaxis and bloody stools
Cardiac Arrhythmias (Cardiac disorders) | 7 (9) | 0 (0)
Other (Volume Overload) (Cardiac disorders) | 1 (1) | 0 (0) — Volume overload
Other (decompensated heart failure) (Cardiac disorders) | 1 (1) | 0 (0) — decompensated heart failure
Right Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
Other (vasodilatory shock periop) (Vascular disorders) | 1 (1) | 0 (0) — vasodilatory shock periop
Device Malfunction-Pump Thrombus-Suspected (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Major Infection - Percutaneous Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Major Infection - Internal Pump Component, Inflow, or Outflow Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Neurological Dysfunction - Ischemic Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Ischemic stroke
Neurological Dysfunction - TIA (Nervous system disorders) | 1 (1) | 0 (0) — TIA
Neurological Dysfunction - Other (Nervous system disorders) | 1 (1) | 0 (0) — focal seizures
Renal Dysfunction - Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Other (New diagnosis of Type II diabetes) (Endocrine disorders) | 0 (0) | 1 (1) — New diagnosis of Type II diabetes

LIMITATIONS AND CAVEATS:
After the 10th patient was enrolled,enrollment was permanently suspended due to a change in NIH funding. Enrollment activity ceased and study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site investigators have the right to independently publish results of their portion of the study conducted at their site 1 year following study conclusion; the site investigator must submit to the DCC for review and comment,a copy of any proposed manuscript resulting from research at least thirty (30) days prior to estimated publication date. If no response is received within thirty (30) days of the date the manuscript was submitted to the DCC, publication may proceed without delay.